CLINICAL TRIAL: NCT05228392
Title: The Effects of Listening to Lullabies and Self-selected Music on Distress and Maternal Attachment in Pregnant Women: A Randomized-controlled Study
Brief Title: The Effects of Listening to Lullabies and Self-selected Music on Distress and Maternal Attachment in Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nazlı Baltacı, Assistant Professor, phD, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 365
Record Dates: First submitted 2022-01-12; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Psychological Distress; Bonding

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- lullaby group (Experimental): For two weeks and 30 minutes every day at home, the lullaby group (LG) only listened to the lullaby record selected by the researcher
  Interventions: Other: listening to music
- multi music group (Experimental): For two weeks and 30 minutes every day at home, the multi-music group (MG) listened to self-selected music from different records presented to them by the researcher.
  Interventions: Other: listening to music
- control group (No Intervention): The control group (CG) only received routine care. This group do not listened to music.

INTERVENTIONS:
Other: listening to music — listening to lullaby or other music types
  Arms: lullaby group; multi music group

SUMMARY:
The purpose of this study is to compare the effects of listening to lullabies and self-selected music at home in reducing the distress experienced in the prenatal period and increasing maternal attachment in pregnant women. This parallel randomized-controlled study was carried out at obstetrics outpatient clinics in Turkey. For two weeks and 30 minutes every day at home, the lullaby group (LG) only listened to the lullaby record selected by the researcher, while the multi-music group (MG) listened to self-selected music from different records presented to them by the researcher. The control group (CG) only received routine care. Prenatal distress and maternal attachment levels were assessed at the beginning and end of the intervention.

DETAILED DESCRIPTION:
Pregnant women may experience distress due to physical and psychosocial changes, and this distress affects the development of maternal attachment negatively. Healthcare professionals are supposed to assess the distress and maternal attachment levels of pregnant women, facilitate their development of positive coping mechanisms, reduce their distress and increase their attachment. In this sense, music interventions may be utilized to improve the physical, emotional and mental health of pregnant women. Based on the information in the literature, it is known that music therapy can be implemented at home, too. In some studies that included music interventions carried out at home, anxiety and stress were reduced, and thus, psychological benefits were facilitated for the pregnancy, labor and postpartum periods. The purpose of this study is to compare the effects of listening to lullabies and self-selected music at home in reducing the distress experienced in the prenatal period and increasing maternal attachment in pregnant women.

This study is an experimental, parallel-group, pretest-posttest randomized-controlled study that was carried out in compliance with the instructions of CONSORT (as given in the CONSORT Checklist 2010). The study was conducted at the obstetrics outpatient clinics of a state hospital located in northern Turkey. The population of the study consisted of healthy pregnant women presenting to the obstetrics outpatient clinics of the hospital where the study was conducted for their pregnancy follow-ups. The sample size was calculated using the G*Power 3.1.9 software. It was determined that each group should include at least 36 pregnant women according to a 95% confidence interval (1-α), an error margin of 0.05, a power rate of 0.95 and an effect size of d=0.87. The pregnant women who were included in the study (n=120) were allocated to the lullaby group (LG) (n=40), the multi-music group (MG) (n=40) or the control group (CG) (n=40) using the simple randomization method. The specialist randomly allocated each participant to one of the intervention groups (LG and MG) or CG using the "QuickCalcs - Graph Pad" computer program.Participants who met the inclusion criteria were included in the groups based on their orders of presenting to the obstetrics outpatient clinics which were randomly distributed.

The data of the study were collected using a Personal Information Form, the Prenatal Distress Questionnaire, and the Maternal Antenatal Attachment Scale. Prenatal distress and attachment levels were assessed at the beginning of the study (pretest) and at the end of the 2-week music intervention/two weeks of routine care (posttest). All data were collected at the hospital when the pregnant women arrived there for their pregnancy follow-ups.

The study included two intervention groups and a control group (CG). The interventions groups were the lullaby group (LG) and the multi-music group (MG). The participants in the control group did not listen to music. They only received the routine care offered to them in their hospital visits.

Music interventions (LG and MG) The participants in LG were instructed to only listen to the recording of lullabies selected by the researcher for two weeks and 30 minutes every day at home. The participants in MG were given records of music consisting of "nature sounds, Western classical music, Turkish classical music (in the acemaşiran mode) and lullabies" that were arranged by the researcher and instructed to listen to select and listen to any of these at home for two weeks and 30 minutes every day.The participants in the music intervention groups were informed about the form and conditions of listening to the given music records at their homes. The music files were sent to the participants via mobile communication applications (e.g., Telegram, WhatsApp) so that they could listen to them on their own phones, and the participants were asked to download/save these files. An instructor at the Musicology department of the university where this study was implemented was consulted regarding these music records. Based on information published in previous studies, a guide for listening to music at home in pregnancy was developed [12,16]. Accordingly, lullabies compatible with a normal heart rate (varying in the range of 60-70 bpm as measured with a metronome) and with a soft melody and other music pieces mentioned above were used. The participants were instructed to use their personal headphones in a quiet and dimly lit room to prevent the effects of ambient sounds while listening to music, adjust the volume of the music to a level that they preferred and was appropriate, empty their bladder and not be hungry. The appropriate implementation of these music interventions at home was checked by the researcher by having phone calls with the participants every day.

Due to the nature of music interventions, the researchers and the participants were not blind to the study protocol. No intervention was made in the routine care and follow-up processes of the participants throughout the study.

Data analysis:

All data were analyzed using the IBM SPSS v.23 (IBM Corp. Armonk, NY, USA) program. The results are presented with descriptive statistics including frequency, percentage, arithmetic mean, standard deviation, median, minimum and maximum values. Chi-squared test was used for the categorical variables, and one-way analysis of variance (ANOVA) or Kruskal Wallis-H test was used for the continuous variables to confirm differences in sociodemographic and obstetrics characteristics between the groups. The mean NuPDQ and MAAS scores of the groups were compared using one-way analysis of variance (ANOVA) and Tukey's test, while intragroup comparisons were made using paired-samples t-test. The level of statistical significance was accepted as p<0.05.

Ethical considerations:

Before starting the study, ethical approval was obtained from the Clinical Research Ethics Committee of the university where the study would be conducted (decision data: 10.06.2021, decision number: 2021/288), and written permission was received from the institution. Additionally, before implementing the data collection instruments, the aim of the study was explained to all participants, and written informed consent was obtained from those who voluntarily agreed to participate.

Limitations There were some limitations in this study. First, as this study was a single-center study, its results cannot be generalized to all healthy pregnant women. Second, as no follow-up was made after the two-week music intervention in the study or in the postpartum period, the long-term effectiveness of having pregnant women listen to lullabies or other music genres could not be analyzed. Third, asking the participants to listen to music at home and checking their compliance over the phone created difficulties in terms of comprehensive implementation in terms of issues such as the duration of the intervention and its implementation conditions.

ELIGIBILITY:
Inclusion Criteria:

* Agreeing to participate in the study
* Being 19 years old or older,
* Being in the third trimester of pregnancy
* Having a singleton pregnancy
* Not having any fetal anomaly
* Being literate
* Using a mobile communication application (e.g., Telegram, WhatsApp)
* Not having a psychiatric disorder
* Being able to communicate in Turkish.

Exclusion Criteria:

* Not agreeing to participate
* Having a risky pregnancy
* Being in the first or second trimester of pregnancy
* Having a multiple pregnancy
* Having a fetal anomaly
* Having a mental, cognitive, psychiatric, auditory or visual disorder or impairment
* Being illiterate
* Not using a mobile communication application (e.g., Telegram, WhatsApp)
* Not being able to communicate in Turkish.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Psychological bonding change | At baseline and at the end of the 2nd week of study, psychological bonding was assessed.
  As assessed by the "Maternal Antenatal Attachment Scale" (MAAS) developed by Condon (1993).Each item of the scale, which consists of a total of 19 items, focuses on the feelings, attitudes and behaviors of the pregnant woman towards her fetus. The minimum and maximum total scores of the scale are 19 and 95. Higher scores show higher levels of prenatal maternal attachment.
Psychological distress change | At baseline and at the end of the 2nd week of study, psychological distress was assessed.
  As assessed by the "Prenatal Distress Questionnaire" (NuPDQ) that was developed by Yali and Lobel (1999). This 3-point Likert-type scale consisting of 17 items in total determines physical and emotional symptoms that could arise in pregnancy, relevant relationships, problems or concerns experienced in issues associated with motherhood, body image and pregnancy. The pregnancy-specific distress experienced in the pregnancy period is scored by summing the scores of the respondent in all items. The minimum and maximum total scores of the scale are 0 and 34. Higher scores are interpreted as higher levels of prenatal distress.

CONTACTS AND LOCATIONS:
Overall Officials: Nazlı Baltacı, phD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Samsun Training and Research Hospital, Obstetrics and Gynecology Clinic, Gynecology and Obstetrics Polyclinics, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Baltaci N, Koc E, Dogan Yuksekol O, Cokyeter B. The Effects of Listening to Lullabies and Self-selected Music on Distress and Maternal Attachment in Pregnant Women: A Randomized Controlled Study. Altern Ther Health Med. 2023 Oct;29(7):46-51. PMID 36399083